CLINICAL TRIAL: NCT03929926
Title: Proactive Outreach and Shared Decision Making to Improve Lung Cancer Screening Rates Among Primary Care Patients
Brief Title: Proactive Outreach and Shared Decision Making in Improving Lung Cancer Screening Rates in Primary Care Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Thomas Jefferson University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 18G.752; JT 13384 (Other: JeffTrial Number)
Record Dates: First submitted 2019-04-24; First posted 2019-04-29 (Actual); Last update posted 2025-05-20 (Actual); Status verified 2025-05

CONDITIONS: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms | interventions — Practice Guidelines as Topic; Standard of Care; Counseling

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Group 1 (usual care) (Active Comparator): receive usual care
  Interventions: Other: Best Practice
- Group II (outreach contact) (Experimental): Patients receive educational materials in the mail about lung cancer screening with a cover letter from their physician. A week later, they receive a phone call from the study staff to assess their eligibility. Eligible and interested patients receive an office visit at the JLCSP for shared decision-making and possible lung cancer screening.
  Interventions: Behavioral: Cancer Educational Materials; Other: Behavioral, Psychological or Informational Intervention
- Group III (outreach + Decision Counseling Program) (Experimental): Patients receive educational materials in the mail about lung cancer screening with a cover letter from their physician. A week later, they receive a phone call from the study staff to assess their eligibility. Patients then undergo a decision counseling session through a semi-structured Decision Counseling Program that includes a review of the mailed educational materials and completion of an interactive exercise intended to clarify personal preference related to screening options (to have LDCT or not to have LDCT). Patients interested in screening schedule an office visit at JLCSP for possible screening or are referred to their primary care physician for consultation.
  Interventions: Behavioral: Cancer Educational Materials; Other: Behavioral, Psychological or Informational Intervention; Other: Counseling

INTERVENTIONS:
Other: Best Practice — receive usual care
  Other Names: standard of care; standard therapy
  Arms: Group 1 (usual care)
Behavioral: Cancer Educational Materials — Receive educational materials via mail
  Arms: Group II (outreach contact); Group III (outreach + Decision Counseling Program)
Other: Behavioral, Psychological or Informational Intervention — Receive shared decision making and lung cancer screening information
  Arms: Group II (outreach contact); Group III (outreach + Decision Counseling Program)
Other: Counseling — Undergo decision counseling session
  Other Names: Counseling intervention
  Arms: Group III (outreach + Decision Counseling Program)

SUMMARY:
This trial studies how well proactive outreach and shared decision making works in improving lung cancer screening rates in primary care patients. Proactive outreach and shared decision making strategies may help to improve the detection of lung cancer at an earlier stage through screening.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To compare the combined intervention group (Outreach Contact Group [OC]/Outreach Contact and Decision Counseling Group [OC-DCP]) versus the control usual care group (UC) with respect to time to screening with low dose computed tomography (LDCT).

SECONDARY OBJECTIVES:

I. To compare the combined intervention (OC/OC-DCP) and usual care (UC) groups with respect to the fraction of patients who are referred/scheduled for screening.

II. To compare the combined intervention (OC/OC-DCP) and usual care (UC) groups with respect to the proportion of the referred/scheduled patients who actually keep their screening appointment.

III. To determine cost of implementing the OC and OC-DCP interventions.

EXPLORATORY OBJECTIVES:

I. To compare the two intervention groups (OC-DCP versus [vs.] OC) on the primary and secondary study endpoints (time to LDCT screening, proportion of patients referred/scheduled for screening, proportion of patients keeping their screening appointments, and cost).

II. To assess the feasibility of patient eligibility review by providers in the OC and OC-DCP arms.

III. To assess the difference in success in identifying eligible patients between arms.

IV. To assess the difference in reaching referred patients between arms.

OUTLINE: Patients are randomized to 1 of 3 groups.

GROUP I (USUAL CARE): Patients receive usual care.

GROUP II (OUTREACH CONTACT): Patients receive educational materials in the mail about lung cancer screening with a cover letter from their physician. A week later, they receive a phone call from the study staff to assess their eligibility. Eligible and interested patients receive an office visit at the Jefferson Lung Cancer Screening Program (JLCSP) for shared decision-making and possible lung cancer screening.

GROUP III (OUTREACH + DECISION COUNSELING PROGRAM): Patients receive educational materials in the mail about lung cancer screening with a cover letter from their physician. A week later, they receive a phone call from the study staff to assess their eligibility. Patients then undergo a decision counseling session through a semi-structured Decision Counseling Program that includes a review of the mailed educational materials and completion of an interactive exercise intended to clarify personal preference related to screening options (to have LDCT or not to have LDCT). Patients interested in screening schedule an office visit at JLCSP for possible screening or are referred to their primary care physician for consultation.

After completion of study, patients are followed up for 90 days.

ELIGIBILITY:
Inclusion Criteria:

* Had a recent office visit with a primary care physician in one of the study practices.
* History of smoking (current or former) in the electronic health record (EHR).

Exclusion Criteria:

* LDCT performed in the 12 months prior to study initiation according to EHR.
* Diagnosis of lung cancer indicated in problem list in the EHR.

Ages: 55 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2355 (Actual)
Dates: Start 2019-06-19 (Actual); Primary Completion 2024-01-01 (Actual); Study Completion 2024-05-01 (Actual)

PRIMARY OUTCOMES:
Time to screening with low dose computed tomography (LDCT) | From the date of randomization to the date of screening (for those screened) or to the date of the review (for those not screened, "censored", assessed at 3 months
  Will be assessed through a review of electronic health records data at the end of the study. The main analysis will compare the combined intervention group and the usual care group (Outreach Contact [OC]/OC-Decision Counseling Program [DCP] versus [vs.] usual care [UC]) with the Kaplan-Meier method and the log-rank test (stratified by practice). Further analyses will rely on Cox proportional hazards regression to explore the difference between OC and OC-DCP groups, as well as differences across practices and patient characteristics (age, gender, race, current vs. former smoking, etc.).

CONTACTS AND LOCATIONS:
Overall Officials: Ronald Myers, Principal Investigator — Sidney Kimmel Cancer Center at Thomas Jefferson University
Locations (1):
- Sidney Kimmel Cancer Center at Thomas Jefferson University, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No